CLINICAL TRIAL: NCT01962896
Title: A Phase II Study of Sirolimus and Erlotinib in Recurrent/Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Theodore Laetsch (Other)
Responsible Party: Sponsor-Investigator, Theodore Laetsch, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTSW-GCT-001
Record Dates: First submitted 2013-09-20; First posted 2013-10-14 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Relapsed / Recurrent Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Erlotinib Hydrochloride; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + sirolimus (Experimental)
  Interventions: Drug: Erlotinib; Drug: Sirolimus

INTERVENTIONS:
Drug: Erlotinib
Drug: Sirolimus

SUMMARY:
The purpose of this study is to find out if the combination of an mTOR inhibitor (sirolimus) with an EGFR inhibitor (erlotinib) is effective at treating relapsed or refractory germ cell tumors, and to find out what the side-effects of this regimen are.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than 12 months and less than 50 years of age at the time of study enrollment.
* Patients must have had histologic verification of an extracranial germ cell tumor that is not a pure mature teratoma.
* Patients must have sufficient tumor tissue available to allow assessment of EGFR and mTOR pathway activation (see Section 5.2.3 for sample requirements)
* Patients must have relapsed or refractory disease following at least two prior cisplatin containing chemotherapy regimens.
* Patients must have measurable disease, documented according to RECIST criteria, or evaluable disease with a standard tumor marker (AFP and/or HCG) greater than 10 times the upper limit of normal.
* Patients must have a Lansky or Karnofsky performance status score of ≥ 50. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age.
* Patients must have a life expectancy of greater than 8 weeks.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy.

  * Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment.
  * Patients must be > 7 days since treatment with hematopoetic growth factors (>14 days for Neulasta).
  * Patients must be >7 days since therapy with a biologic agent and beyond the period for which adverse events of the biologic agent are known to occur if longer.
  * Patients must be >3 half-lives since therapy with a monoclonal antibody.
  * Patients must be >42 days since completion of any immunotherapy (i.e. tumor vaccines).
  * Patients must be greater than 2 weeks since most recent palliative XRT and greater than 6 weeks since substantial bone marrow irradiation.
  * Patients must be greater than 8 weeks since prior stem cell transplant or infusion and without evidence of active graft vs. host disease.
* Adequate bone marrow function defined as:

  * Peripheral absolute neutrophil count (ANC) of at least 1,000/ L
  * Platelet count of at least 100,000/ L (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
  * Hemoglobin 8.0 g/dL (may receive RBC transfusions).
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope GFR 70 mL/min/1.73 m2 or
  * Maximum serum creatinine (mg/dL) based on age/gender
* Adequate liver function defined as:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) ≤ 2.5 x ULN (for the purpose of this study, the ULN for SGPT is 45 U/L)
  * Serum albumin ≥ 2 g/dL.
* Adequate central nervous system function defined as:

  o Patients with seizure disorder may be enrolled if receiving non-enzyme inducing anticonvulsants and well controlled.
* Serum cholesterol levels must be less than Grade 2 (< 300 mg/dL), and serum triglyceride levels must be less than Grade 2 (< 2.5 x ULN).

Exclusion Criteria:

* Patients with active brain metastases are not eligible as lethal intratumoral hemorrhages have been reported with erlotinib therapy. Patients with brain metastases that have been treated and stable for > 30 days following treatment will be eligible.
* Patients who are pregnant or breast feeding will not be entered into the study as erlotinib is teratogenic. Pregnancy tests must be obtained in females who are post-menarchal. Post-menarchal females with HCG secreting tumors will be excluded as pregnancy can't be excluded. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of the study.
* Concomitant medications

  * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
  * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
  * Anticonvulsants: Patients who are receiving enzyme-inducing anticonvulsants are not eligible (see Appendix 1 for a list of enzyme- inducing anticonvulsants).
  * Anticoagulants: Use of warfarin is not allowed while on study. Patients already on warfarin should use alternative anticoagulants while on this study. Warfarin must not have been administered within 7 days of enrollment.
  * Smoking: Smoking induces CYP3A4/5 enzymes and decreases exposure to sirolimus and erlotinib. Thus, patients must not smoke for 10 days prior to enrollment and for the duration of therapy.
* Infection: Patients who have an uncontrolled infection are not eligible.
* Drug interactions: Sirolimus and erlotinib are primarily metabolized by the CYP3A4/5 enzymes. Drug exposure is substantially effected by CYP inhibitors (increased exposure) and inducers (decreased exposure). Thus, concomitant administration of strong CYP3A4/5 inhibitors or inducers is prohibited while on therapy. See Appendix 1 for a list of these medications. Patients must not have received these medications for a minimum of 10 days prior to enrollment.
* Patients who have received prior therapy targeting EGFR with small molecule tyrosine kinase inhibitors or monoclonal antibodies are NOT eligible.
* Prior treatment with mTOR or TORC1/2 inhibitors (eg, rapamycin, temsirolimus, everolimus, sirolimus) is NOT allowed.
* Patients who have had major surgery within 3 weeks prior to enrollment are not eligible. Procedures such as placement of a central vascular catheter, or limited tumor biopsy, are not considered major surgery.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2018-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center/Children's Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib + Sirolimus: Erlotinib 85 mg/m2, max of 150 mg, was administered orally once daily continuously. Intrapatient dose escalation and de-escalation rules provided in the protocol.
  Sirolimus was started at a dose of 1 mg/m2, maximum 2mg, orally once daily continuously. The dose of sirolimus was be adjusted at least weekly to obtain a goal trough level of 10-15ng/mL.
Period: Overall Study
Arm/Group | Erlotinib + Sirolimus
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib + Sirolimus: Erlotinib
  Sirolimus
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The PFR, Defined as the Proportion of Patients With Refractory Germ Cell Tumors Free of Objective Disease Progression After 4 Cycles (16 Weeks) of Therapy With Erlotinib and Sirolimus
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Progressive Disease (PD), >= 20% increase in the sum of the longest diameter of target lesions or the development of any new lesions
Time Frame: 16 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 4
percentage of patients | 0

2. Primary Outcome: The Toxicities of the Combination of Sirolimus and Erlotinib Administered on This Schedule.
Description: The number of patients with drug related grade III, IV, or V adverse events according to the Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 4
Participants
  CTCAE v4 grade 3 AE | 2
  CTCAE v4 grade 4 AE | 0
  CTCAE v4 grade 5 AE | 0
  No CTCAE v4 Grade >2 AE | 2

3. Secondary Outcome: The Incidence of EGFR and mTOR Pathway Activation in Banked Tumor Specimens.
Time Frame: 3 years
Population: Analysis was not performed as the study was terminated early without sufficient enrollment to analyze this objective.
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 0

4. Secondary Outcome: The Progression-free Interval (PFI) for Patients With Germ Cell Tumors With and Without Evidence of EGFR/mTOR Pathway Activation With This Drug Combination.
Time Frame: 3 years
Population: Analysis was not performed as the study was terminated early without sufficient enrollment to analyze this objective.
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from enrollment until the patient came off study, up to 2 years
Arm/Group | Erlotinib + Sirolimus
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Sirolimus (N=4)
Rash (Skin and subcutaneous tissue disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 2
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2
Alanine aminotransferrase increased (Hepatobiliary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT01962896/Prot_SAP_000.pdf